CLINICAL TRIAL: NCT02735733
Title: Does Cold Saline Used to Inflate a Balloon Tamponade Catheter More Significantly Reduce Blood Loss From Postpartum Hemorrhage Than Room Temperature Saline?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study never started
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Supportive Care
Other Study IDs: 016-092
Record Dates: First submitted 2016-04-07; First posted 2016-04-13 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Room temperature arm (Active Comparator): Intervention: The balloon catheter will be placed through the vagina into the uterus and inflated using normal saline at room temperature.
  Interventions: Device: Cold Bakri Balloon
- Cold arm (Experimental): Intervention: The balloon catheter will be placed through the vagina into the uterus and inflated using normal saline at approximately 32 degrees F for the study group.
  Interventions: Device: Cold Bakri Balloon

INTERVENTIONS:
Device: Cold Bakri Balloon — In the room temperature arm, the bakri balloon will be inserted through the vagina and placed inside the uterus and filled with room temperature saline. In the cold arm, the same intervention will performed, however, the bakri balloon will be filled with cold saline at 32 degrees Fahrenheit.

SUMMARY:
To determine if a balloon tamponade catheter filled with cold saline is more effective than a catheter filled with room temperature saline in controlling post partum hemorrhage.

DETAILED DESCRIPTION:
When post partum hemorrhage occurs one mode of therapy is to place a balloon tamponade catheter into the uterus to compress the bleeding vessels. When this mode of therapy has been chosen by the attending physician the patient will be randomized to either the room temperature arm (control) or the cold arm (study). The balloon catheter is placed through the vagina into the uterus and inflated using normal saline; room temperature for the control group and approximately 32 degrees F for the study group. Traction is placed on the catheter to tamponade the vessels in the lower uterine segment. Blood from the uterus passes through a central lumen of the balloon and will be collected and measured. Total measured blood loss for each group will be compared.

ELIGIBILITY:
Inclusion Criteria:

* women 18-45 years old who have just delivered they baby vaginally who now have uncontrolled bleeding from their uteri

Exclusion Criteria:

* anyone outside of the specified age group
* anyone who declines to participate in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-04-08 (Actual); Study Completion 2016-04-08 (Actual)

PRIMARY OUTCOMES:
Total measured blood loss | time frame is approximately 24 hours, until the balloon catheter is removed from the uterus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kellie FJ, Wandabwa JN, Mousa HA, Weeks AD. Mechanical and surgical interventions for treating primary postpartum haemorrhage. Cochrane Database Syst Rev. 2020 Jul 1;7(7):CD013663. doi: 10.1002/14651858.CD013663. PMID 32609374